CLINICAL TRIAL: NCT03865537
Title: Cold Endoscopic Resection of Large Colorectal Polyps: A Randomized Trial
Brief Title: Cold Snare Endoscopic Mucosal Resection Trial
Acronym: LPS-II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Dartmouth College (Other); Steris (Unknown); Cosmo Pharmaceuticals (Unknown)
Responsible Party: Principal Investigator, Dr. Heiko Pohl, Associate Professor or Medicine, White River Junction Veterans Affairs Medical Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 119681
Record Dates: First submitted 2019-03-03; First posted 2019-03-07 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Colonic Polyp; Colonoscopy; Complication; Recurrence
MeSH Terms: conditions — Colonic Polyps; Recurrence | interventions — SIC-8000

STUDY DESIGN:
Intervention Model Description: 2 x 2 randomized trial.
  First randomization: Among half of patients with a large polyp will be removed by electrocautery ("hot") snare resection, and the other half will have their polyp removed by snare resection without electrocautery ("cold").
  Second randomization: Among half of patients the large polyp will by lifted (submucosal injection before resection) with Eleview; among the other by Placebo (Normal Saline with Methylene Blue).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization 1 (Cold vs. hot snare group): Masking only of participants Randomization 2 (Eleview vs Placebo): Masking of all checked above
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cold snare & Eleview injection (Experimental): Polyp resection without electrocautery (cold snare EMR), and initial submucosal injection with Eleview
  Interventions: Procedure: Cold snare EMR; Procedure: Eleview injection
- Cold Snare & Placebo injection (Experimental): Polyp resection without electrocautery (cold snare EMR), and initial submucosal injection with Placebo
  Interventions: Procedure: Cold snare EMR; Procedure: Placebo injection
- Hot snare & Eleview injection (Active Comparator): Polyp resection with electrocautery (hot snare EMR), and initial submucosal injection with Eleview
  Interventions: Procedure: Hot snare EMR; Procedure: Eleview injection
- Hot snare & Placebo injection (Active Comparator): Polyp resection with electrocautery (hot snare EMR), and initial submucosal injection with Placebo
  Interventions: Procedure: Hot snare EMR; Procedure: Placebo injection

INTERVENTIONS:
Procedure: Cold snare EMR — Participants will have their large polyp removed without electrocautery
  Arms: Cold Snare & Placebo injection; Cold snare & Eleview injection
Procedure: Hot snare EMR — Participants will have their large polyp removed with electrocautery
  Arms: Hot snare & Eleview injection; Hot snare & Placebo injection
Procedure: Eleview injection — Participants will have their polyp submucosally injected with Eleview
  Arms: Cold snare & Eleview injection; Hot snare & Eleview injection
Procedure: Placebo injection — Participants will have their polyp submucosally injected with placebo
  Arms: Cold Snare & Placebo injection; Hot snare & Placebo injection

SUMMARY:
This study compares different approaches to endoscopic mucosal resection (EMR) of large non-pedunculated colorectal polyps (≥20mm) in a 2 x 2 randomized design. The first randomization will assign half of patients to polyp resection with electrocautery ("hot" snare EMR) and half of patient to polyp resection without electrocautery ("cold" snare EMR). The second randomization will assign half of patients to polyp removal using Eleview as the submucosal injection agent, and the other half using placebo (normal saline with methylene blue) as the submucosal injection agent.

DETAILED DESCRIPTION:
Electrocautery, or hot snare resection has long been considered the standard approach to polyp resection. A major limitation is a 5 to 10% risk of major adverse events. Recent studies suggest that snare resection without electrocautery - so-called cold snare EMR - may be safer than hot snare EMR. The concern with cold snare resection is a potentially lower efficacy, because cold snare resection requires the removal of a large polyp in smaller and greater number of pieces than with hot snare resection. This may lengthen procedure time and increase the risk of incomplete resection.

Furthermore, there is uncertainty about the optimal injection solution for lifting of the polyp prior to resection. Normal saline with methylene blue as the contrast agent is frequently used, but is limited by fast dissipation of the polyp lift. Eleview is a newly approved viscous solution (that contains methylene blue), which provides a longer polyp lift than normal saline. It is unclear how these two solutions compare with respect to resection efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Any patient ≥18 who presents for a colonoscopy and who does not have criteria for exclusion
* Patients with a ≥20mm non-pedunculated colorectal polyp

Exclusion Criteria:

* Pedunculated polyps (as defined by Paris Classification type Ip)
* Suspected adenocarcinoma with deep submucosal invasion
* Patients with ulcerated depressed lesions (as defined by Paris Classification type III) or confirmed adenocarcinoma
* Patients with inflammatory bowel disease
* Patients who are receiving an emergency colonoscopy
* Poor general health (ASA class>3)
* Patients with coagulopathy with an elevated INR ≥1.5, or platelets <50
* Inadequate bowel preparation (Boston Bowel Prep Scale, total score ≤2)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 990 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Severe Adverse Events | up to 30 days following the procedure
  Aggregate of all severe adverse events that occur at the time of the colonoscopy with resection of the large polyp or following the procedure

SECONDARY OUTCOMES:
Subcategories of severe adverse events | during the procedure and up to 30 days following the procedure
  Bleeding, post-polypectomy syndrome, perforation, abdominal pain
Performance submucosal injectate | immediately following polyp resection during the colonoscopy
  Injection performance
Volume of submucosal injectate | immediately following polyp resection during the colonoscopy
  volume of injection
Efficacy of submucosal injectate | immediately following polyp resection during the colonoscopy
  Sidney index
Completeness of polyp resection | immediately following polyp resection during the colonoscopy
  Complete polyp removal is defined as removal of all visible polyp tissue at the end of the EMR, as assessed by the endoscopist.
Intraprocedural bleeding | at the time of polyp resection
  bleeding that requires endoscopic intervention to stop the bleeding
Polyp recurrence | at surveillance colonoscopies up to 5 years following the initial polyp resection
  Presence of biopsy proven neoplastic polyp tissue at the EMR resection site at surveillance colonoscopy following complete polyp resection
Crossover from cold to hot snare | at the time of polyp resection
  Proportion of polyps in the cold snare group that could not be removed by cold snare and were removed by hot snare, categorized by size and morphology subtypes of polyps

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Pohl, MD, Study Chair — White River Junction VAMC, Geisel School of Medicine at Dartmouth
Locations (1):
- White River Junction VAMC, White River Junction, Vermont, United States

REFERENCES:
- [Derived] Pohl H, Rex DK, Barber J, Moyer MT, Elmunzer BJ, Rastogi A, Gordon SR, Zolotarevsky E, Levenick JM, Aslanian HR, Elatrache M, von Renteln D, Wallace MB, Brahmbhatt B, Keswani RN, Kumta NA, Pleskow DK, Smith ZL, Abu Ghanimeh MK, Simmer S, Sanaei O, Mackenzie TA, Piraka C. Cold snare endoscopic resection for large colon polyps: a randomised trial. Gut. 2025 Oct 8;74(11):1804-1813. doi: 10.1136/gutjnl-2025-335075. PMID 40393701